CLINICAL TRIAL: NCT07062965
Title: An Interventional, Open-Label, Randomized, Multicenter, Phase 3 Study of PF-07248144 Plus Fulvestrant Compared to Investigator's Choice of Therapy in Adult Participants With Hormone Receptor-Positive, HER2-Negative Advanced/Metastatic Breast Cancer Whose Disease Progressed After Prior CDK4/6 Inhibitor-based Therapy
Brief Title: A Study to Learn About the Study Medicine Called PF-07248144 in Combination With Fulvestrant in People With HR-positive, HER2-negative Advanced or Metastatic Breast Cancer Who Progressed After a Prior Line of Treatment.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4551002; 2025-520566-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Locally advanced or metastatic breast cancer; Estrogen receptor positive [ER(+)]; Progesterone receptor positive [PR(+)]; Human epidermal growth factor receptor 2 negative [HER2(-)]; ER(+)/HER2(-); PR(+)/HER2(-); HR(+)/HER2(-); Advanced Breast Cancer; Breast tumor; Breast cancer; Everolimus; Exemestane; Fulvestrant; Metastatic breast cancer; Endocrine Therapy; Hormone Therapy; Hormone positive breast cancer; Recurrent breast cancer; HR+; HER2-negative; Relapse; Recurrent; Second line treatment; Third line treatment; Left Sided Breast Cancer; Right Sided Breast Cancer; Unilateral Breast Cancer; Cancer of the Breast; CDK4/6i; CDK4/6i-based Therapy; Bilateral Breast Cancer; Progression After CDK4/6i-based therapy
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Unilateral Breast Neoplasms | interventions — Fulvestrant; Everolimus; exemestane

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned into 1 of 2 groups in parallel for the entire duration of the study. The experimental arm will receive PF-07248144 and fulvestrant (Arm A) while the comparator arm will receive everolimus in combination with the study doctor's choice of endocrine therapy (exemestane or fulvestrant; Arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: PF-07248144 plus fulvestrant (Experimental): PF-07248144 tablet taken by mouth plus fulvestrant taken as a shot into the muscle.
  Interventions: Drug: PF-07248144; Drug: Fulvestrant
- Arm B: everolimus plus ET (Active Comparator): Everolimus tablet taken by mouth plus investigator's choice of endocrine therapy of exemestane tablet taken by mouth or fulvestrant taken as a shot into the muscle.
  Interventions: Drug: Fulvestrant; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: PF-07248144 — KAT6 inhibitor
  Arms: Arm A: PF-07248144 plus fulvestrant
Drug: Fulvestrant — Endocrine therapy
Drug: Everolimus — mTOR inhibitor
  Arms: Arm B: everolimus plus ET
Drug: Exemestane — Endocrine therapy
  Arms: Arm B: everolimus plus ET

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine PF-07248144 when given along with fulvestrant for the possible treatment of HR-positive, HER2-negative advanced or metastatic breast cancer.

HR-positive breast cancer cells have proteins on their surface called receptors that bind to hormones like estrogen and progesterone (female sex hormones). These hormones can promote the growth of cancer cells.

HER2-negative describes cells that have a small amount or none of a protein called HER2 on their surface. In normal cells, HER2 helps control cell growth. Cancer cells that are HER2-negative may grow more slowly and are less likely to recur (come back) or spread to other parts of the body than cancer cells that have a large amount of HER2 on their surface.

Advanced cancer is a term that is often used to describe cancer that is unlikely to be cured.

Metastatic cancer is the type where the cancer cells spread from one part of the body to another.

This study is seeking for participants whose breast cancer has gotten worsen after receiving cyclin dependent kinase (CDK) 4/6 inhibitor-based therapy.

Half of participants in this study will receive their usual study treatment, everolimus with endocrine therapy (either exemestane or fulvestrant) for HR-positive/HER2-negative advanced or metastatic breast cancer (A/mBC). The study doctor will discuss which hormone therapy is right for the participant before treatment begins.

PF-07248144 is a tablet that will be taken by mouth at home every day in a 28-day cycle. Fulvestrant will be given as two injections (one injection in the buttock) at visits to the study clinic. Everolimus and exemestane are also tablets and will be taken by mouth at home every day in a 28-day cycle.

The study will compare the experiences of people receiving PF-07248144 in combination with fulvestrant to those of the people who do not. This will help see if PF-07248144 in combination with fulvestrant is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HR-positive HER2-negative breast cancer with evidence of locally advanced or metastatic disease, which is not amenable to surgical resection or radiation therapy with curative intent.
* Prior CDK4/6 inhibitor therapy in combination with endocrine therapy in advance metastatic setting or in adjuvant setting with documented progression during or within 12 months after the last dose of CDK4/6i.
* Participants are eligible if they previously received CDK4/6i or ET as a monotherapy, or in combination for rechallenge therapy in the advance or metastatic setting; have received prior therapy targeting estrogen receptor 1 (ESR1) or breast cancer gene (BRCA)1/2.
* Measurable disease evaluable per Response Evaluation Criterion in Solid Tumors (RECIST) v.1.1 or non-measurable bone-only disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.

Exclusion Criteria:

* Documented detectable PIK3CA/AKT1/PTEN alterations in tissue
* Received greater than two prior lines of systemic therapy in the advance or metastatic setting
* Had received any prior chemotherapy, including antibody drug conjugates (ADCs), in advance or metastatic setting. Participants who have previously received chemotherapy in the (neo)adjuvant setting are not excluded from the study.
* Any medical or psychiatric condition that may increase the risk of study participation or make the participant inappropriate for the study.
* Renal impairment, hepatic dysfunction, or hematologic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2030-11-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as determined by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From the date of randomization until disease progression or death due to any cause (up to approximately 2 years)

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of randomization until death due to any cause (up to approximately 5 years).
Number of Participants with Objective Response (OR) by BICR | From the date of randomization until disease progression or death due to any cause (up to approximately 2 years)
Duration of Response (DoR) as defined by BICR | From the date of the first objective (PR or CR) response (every 8 weeks during the first 48 weeks and then every 12 week) up to approximately 2 years.
Number of Participants With Clinical Benefit Response (CBR) by BICR | From randomization date (every 8 weeks during the first 48 weeks and then every 12 weeks) up to approximately 2 years.
Number or Patients with Adverse Events (AEs) by Type | From screening until 28 days after the last dose, to approximately 5 years
Number or Patients with AEs by Incidence | From screening until 28 days after the last dose, to approximately 5 years
Number or Patients with AEs by Seriousness | From screening until 28 days after the last dose, to approximately 5 years
Number or Patients with AEs by relationship to study interventions | From screening until 28 days after the last dose, to approximately 5 years
Number of Participants With Abnormal Electrocardiogram (ECG; Arm A and B) | From screening until 28 days after the last dose, to approximately 5 years
Number of Participants With Increase From Baseline in Corrected QT (QTc) Interval (Arm A only) | 0h pre-dose on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, and Cycle 3 Day 1; additional 4 hrs post dose on Cycle 1 Day 15 and Cycle 2 Day 1
  The study includes a QTc sub-study in approximately 40 participants in Arm A enrolled at selected sites which will evaluate the effect of PF-07248144 on QTc interval via collection of triplicate ECGs (central reading) time-matched with pharmacokinetic (PK) draws.
Number of Participants With Laboratory Test Abnormalities | From screening until 28 days after the last dose, to approximately 5 years
Ctrough of PF-07248144 | Cycle 1 (Day 1), Cycle 1 (Day 15), Cycle 2 (Day 1), and Cycles 3, 5, and 7 (Day 1) only. Each Cycle is 28 days
  Ctrough was defined as pre-dose serum concentration during multiple dosing and observed directly from data.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (148):
- United States (58):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Goodyear, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - Los Angeles Cancer Network - Anaheim, Anaheim, California
  - Los Angeles Cancer Network - Fountain Valley, Fountain Valley, California
  - Los Angeles Cancer Network - (Admin Only / Central IDS) - No Patients, Glendale, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Los Angeles Cancer Network - Van Nuys, Los Angeles, California
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Stanford Cancer Center, Palo Alto, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Smilow Cancer Hospital - Derby, Derby, Connecticut
  - Smilow Cancer Hospital - Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital - Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital - Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Hospital - Yale New Haven Health, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital - North Haven, North Haven, Connecticut
  - Smilow Cancer Hospital - Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital - Torrington, Torrington, Connecticut
  - Smilow Cancer Hospital - Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital - Waterbury, Waterbury, Connecticut
  - Smilow Cancer Hospital - Waterford, Waterford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Summit Cancer Care, PC, Savannah, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Prime Saint Francis-Infusion Services Evanston, Evanston, Illinois
  - Memorial Hospital., Shiloh, Illinois
  - Siteman Cancer Center - Shiloh, Shiloh, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Prime Saint Francis-Infusion Services Skokie, Skokie, Illinois
  - Mercy Medical Center - Baltimore, Baltimore, Maryland
  - The Cancer & Hematology Centers, Big Rapids, Michigan
  - The Cancer & Hematology Centers, Grand Rapids, Michigan
  - The Cancer & Hematology Centers, Holland, Michigan
  - The Cancer & Hematology Centers, Norton Shores, Michigan
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - MD Anderson The Woodlands, Conroe, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
- Australia (4):
  - Cancer Research SA Pty Ltd, Adelaide, South Australia
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Western Health-Sunshine & Footscray Hospitals, St Albans, Victoria
- Belgium (4):
  - Algemeen Ziekenhuis klina, Brasschaat, Antwerpen
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - UZ Leuven, Leuven, Vlaams-brabant
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-vlaanderen
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Serdikamed EOOD, Sofia, Sofia (stolitsa)
  - Complex Oncology Center - Burgas, Burgas
  - Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Complex Oncology Center - Shumen, Shumen
  - MHAT for Women's Health Nadezhda, Sofia
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval, Hôpital du Saint-Sacrement, Québec, Quebec
- China (9):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - The 2nd Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice v Motole, Prague, Praha 5
  - Fakultni nemocnice Bulovka, Prague, Praha 8
- Docrates Syöpäsairaala, Helsinki, Uusimaa, Finland
- Greece (4):
  - IASO General Clinic, Athens, Attica
  - Hygeia Hospital, Marousi, Attikí
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
- India (5):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Artemis hospital, Gurugram, Haryana
  - Spandana Oncology Centre (SOC), Bengaluru, Karnataka
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Italy (2):
  - Azienda USL Toscana Nord Ovest_Ospedale Civile di Livorno, Livorno, Tuscany
  - Istituto Europeo di Oncologia IRCCS, Milan
- Japan (15):
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Tokai University Hospital, Isehara, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Japan Institute for Health Security National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjyuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - Okayama University Hospital, Okayama
  - Showa Medical University Hospital, Tokyo
- Netherlands (2):
  - Tergooi MC, Hilversum, North Holland
  - St. Antonius Ziekenhuis, locatie Utrecht, Utrecht
- Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship, Poland
- Ad-Vance Medical Research, Ponce, Puerto Rico
- Slovakia (5):
  - Onkologicky Ustav sv. Alzbety, Bratislava, Bratislava Region
  - Nemocnica s poliklinikou Stefana Kukuru Michalovce a.s., Michalovce, Košice Region
  - Nemocnica AGEL Komarno, Komárno, Nitra Region
  - Narodny onkologicky ustav, Bratislava
  - Nemocnica Bory, a.s., Bratislava
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Kyǒnggi-do
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu, Seoul-teukbyeolsi [seoul]
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-kwangyǒkshi
- Spain (3):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario de Jaen, Jaén
- Sweden (2):
  - Södersjukhuset, Stockholm, Stockholms LÄN [se-01]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands LÄN [se-14]
- Taiwan (6):
  - Chi Mei Medical Center, Tainan, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4551002